CLINICAL TRIAL: NCT04461639
Title: Observational Study Evaluating Long-term Safety of Real-world Treatment With Damoctocog Alfa Pegol in Previously Treated Patients With Hemophilia A
Brief Title: Study to Learn More About the Safety of Drug Jivi Over a Long Period of Time in Previously Treated Patients With Hemophilia A (Bleeding Disorder Resulting From a Lack of FVIII) Who Are Receiving Jivi Regularly at Their Treating Doctors to Prevent Bleeding
Acronym: HA-SAFE
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20904
Record Dates: First submitted 2020-06-18; First posted 2020-07-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Damoctocog alfa pegol: Participants with hemophilia A received damoctocog alfa pegol as prophylaxis treatment prescribed by the physician as part of normal clinical practice.
  Interventions: Drug: Damoctocog alfa pegol (Jivi, BAY94-9027)

INTERVENTIONS:
Drug: Damoctocog alfa pegol (Jivi, BAY94-9027) — Different prophylaxis regimens with damoctocog alfa pegol following approved local labels or any other regimen prescribed by the physician as part of normal clinical practice

SUMMARY:
In this observational study researchers want to learn more about the safety of drug Jivi over a long period of time. Jivi (generic name: Damoctocog alfa pegol) is an approved blood clotting Factor VIII (FVIII) medication for the treatment of hemophilia A (bleeding disorder resulting from a lack of FVIII). It is manufactured via recombinant technology and has an extended half-live, i.e. it will stay longer in the body than other FVIII products. Therefore Jivi acts longer in the body which reduces the frequency of drug injections. This study will enroll previously treated patients with hemophilia A who are receiving Jivi regularly at their treating doctors to prevent bleeding. Observation for each patient will last for at least 4 years, and medical data will be collected during patients' routine visits at their treating doctors.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent/assent will be obtained before any study-related activities
* PTPs with hemophilia A assigned to Jivi prophylaxis treatment
* Negative FVIII inhibitor test before study entry
* Decision to initiate treatment with commercially available Jivi has been made by the treating physician before and independently from the decision to include the patient in this study

Exclusion Criteria:

* Known or suspected contraindications to Jivi or related products
* Mental incapacity, unwillingness or other barriers precluding adequate understanding or cooperation
* Participation in an investigational program with interventions outside of routine clinical practice

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All previously treated patients (PTPs) with hemophilia A receiving prophylaxis with damoctocog alfa pegol will be eligible to be enrolled in the study. Indications and contra-indications according to the local market authorization will be carefully considered
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with safety events | At least 4 years
Duration of safety events | At least 4 years
Number of participants with safety events leading to a change of treatment | At least 4 years
Number of participants with safety events per intensity | At least 4 years
  The maximum intensity of each safety event should be assigned to one of the following categories: mild, moderate or severe
Number of participants with safety events with outcome of death | At least 4 years
Number of participants with safety events related to inhibitor development | At least 4 years

SECONDARY OUTCOMES:
Number of adverse reactions (ARs) that are defined within the system organ classes nervous system and psychiatric disorders | At least 4 years
Number of adverse reactions (ARs) related to hepatic or renal function | At least 4 years
Change from baseline in creatinine | At least 4 years
Change from baseline in estimated glomerular filtration rate (eGFR) | At least 4 years
Change from baseline in alanine transaminase (ALT) | At least 4 years
Change from baseline in aspartate aminotransferase (AST) | At least 4 years
Change from baseline in bilirubin | At least 4 years
Testing for PEG plasma levels (baseline and end of study) | At least 4 years
  PEG (Polyethylene Glycol)-plasma levels at baseline and end of study will be analyzed only if PEG-plasma levels were collected in local routine clinical practice at the investigator's discretion.
Number of patients with abnormal findings as assessed by neurological examination | At least 4 years

CONTACTS AND LOCATIONS:
Locations (6):
- Many Locations, Multiple Locations, Austria
- Many Locations, Multiple Locations, Germany
- Many Locations, Multiple Locations, Greece
- Many Locations, Multiple Locations, Italy
- Many Locations, Multiple Locations, Slovenia
- Many Locations, Multiple Locations, Spain

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.